CLINICAL TRIAL: NCT02787733
Title: Establishing the Effect of Long-term Orange Peel Extract Supplementation on Exercise Performance and Recovery
Brief Title: The Effect of an Orange Peel Extract on Exercise Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioactor (Other)
Collaborators: InnoSportNL (Other)
Responsible Party: Sponsor-Investigator, Bioactor, BioActorBV, Maastricht University Medical Center
Organization: Maastricht University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: WU-PER-001
Record Dates: First submitted 2016-05-24; First posted 2016-06-01 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Exercise Recovery and Endurance
Keywords: performance; recovery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Citrus flavonoid (Experimental): Citrus peel extract containing >90% flavonoids
  Interventions: Dietary Supplement: Citrus flavonoid
- Placebo (Placebo Comparator): Identical looking placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Citrus flavonoid — Daily dose of 500mg divided over two capsules
  Arms: Citrus flavonoid
Dietary Supplement: Placebo — Daily dose of 500mg divided over two capsules
  Arms: Placebo

SUMMARY:
Rationale: Numerous studies have shown the positive effect of a healthy diet and regular moderate exercise. Although, exercise has also been correlated with an increase in reactive oxygen species (ROS) production and a higher incidence of injury. ROS production seems to induce muscle damage, which reduces muscle performance and induces fatigue. Increasing muscle recovery could be an effective way to increase exercise performance. Several food ingredients have been of growing interest due to their specific functioning on the human body. Citrus flavonoids are abundantly available in citrus fruits. Prior studies show a positive effect of citrus flavonoids on endothelial function, by promoting vasodilation. In addition it has a positive effect on the nitric oxide (NO) synthesis, a known compound in regulating endothelial response. This capacity of citrus flavonoids could be useful in stimulating performance and recovery after exercise. Additionally, the ability of scavenging ROS could reduce muscle damage caused by exercise induced oxidative damage.

Objective: Determine the 4-week effect of daily citrus flavonoid supplementation on exercise recovery and performance.

Study design: Randomized, double-blind, placebo-controlled study with parallel design, in which 40 subjects engage in three exercise sessions. The sessions will be subdivided into a pre-test and test 1 and 2. Between test 1 and 2, participants receive daily for 4 weeks citrus flavonoid supplement or a placebo. Each day, subjects should consume 2 capsules each morning, containing in total 500 mg of citrus flavonoids or 500 mg placebo.

Study population: The subjects will be healthy normal weight trained males, with an age of 18 - 25. Additionally, subjects are non-smokers and free of a medication.

Intervention: Participants will be randomly placed in either the citrus flavonoid or placebo group. Participants will be instructed to ingest 2 capsules each morning for 4 consecutive weeks. Each capsule equals to 250 mg of citrus flavonoids or cellulose in case of the placebo treatment.

Main study parameters/endpoints: The main study parameter is the average amount of work load produced during the 10-minute time trail test. In addition, oxygen per minute will be determined as well as the heart rate. Finally, for each test, the subjective rating of perceived exertion (RPE) will be determined during the pre-test and test 1 and 2 by using a Borg scale.

ELIGIBILITY:
Inclusion Criteria:

* Trained participants, defined as engaging at least 3 times a week in moderate to high physical activity for a minimum of 30 minutes
* Non-smoking, defined as no smoking for the last 6 months
* Participants are capable and willing to give written informed consent voluntarily after receiving detailed information from the researchers

Exclusion Criteria:

* Cardiovascular complications
* Extreme BMI (i.e. lower than 18 or higher than 30)
* Use of medication
* Use of antioxidants, minerals and vitamin supplements available in pharmacies, drugstores, food markets or in alternative medicine
* Abuse of products; alcohol (> 20 alcoholic consumptions per week) and drugs
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator) in the 180 days prior to the study
* Failure to comply prohibited intake of hesperidin containing food products during study period. A list with forbidden food products will be provided to participant
* History of any side effects towards the intake of flavonoids or citrus fruits

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Average force output (Watts) in endurance cycling exercise after pre-exhaustive exercise | 4 week
  Average force output is measured through a cycle ergometer

SECONDARY OUTCOMES:
Maximum oxygen uptake (ml/kg/min) in endurance cycling exercise after pre-exhaustive exercise | 4 weeks
  Maximum oxygen uptake is measured through an oxygen mask

CONTACTS AND LOCATIONS:
Overall Officials: Bouke Salden, Drs., Principal Investigator — BioActor
Locations (1):
- InnoSportLab Papendal, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided